CLINICAL TRIAL: NCT00754910
Title: Immunobiology of Photodynamic Therapy in Lung Cancer Patients
Brief Title: Photodynamic Therapy Using Porfimer Sodium in Treating Patients With Non-Small Cell Lung Cancer And Bronchial Disease
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Susan Moffatt-Bruce, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-07115; NCI-2011-03195 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Dihematoporphyrin Ether; Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Patients receive porfimer sodium IV over 3-5 minutes and undergo irradiation with red light 48 hours later. Patients receive 2 more treatments at 2-day intervals.
  Interventions: Drug: porfimer sodium; Procedure: bronchoscopy

INTERVENTIONS:
Drug: porfimer sodium — Given IV
Procedure: bronchoscopy — Patients undergo bronchoscopy

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed. This may be effective against non-small cell lung cancer.

PURPOSE: This clinical trial is studying how well photodynamic therapy using porfimer sodium works in treating patients with non-small cell lung cancer and bronchial disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test the hypothesis that the immune response in non-small cell lung cancer patients treated with photodynamic therapy (PDT) is T cell mediated.

Secondary

* To test the hypothesis that PDT potentially affects survival rates in these patients.
* To test the hypothesis that T lymphocytes mediate an immune response that affects survival in PDT treated patients.

OUTLINE: Patients deemed suitable for photodynamic therapy (PDT) are offered PDT. Patients are divided into 2 groups according to whether or not they receive PDT. All patients are referred to radiation and medical oncology for standard of care adjuvant therapy (beginning after completion of this study).

* Group 1 (PDT): Patients receive porfimer sodium IV over 3-5 minutes and undergo irradiation with red light 48 hours later. Patients receive 2 more treatments at 2-day intervals.
* Group 2 (non-PDT): Patients undergo a baseline bronchoscopy and a repeat bronchoscopy at 4 weeks.

Blood sample, bronchoalveolar lavage fluid, and tumor tissue are collected after each treatment (group 1) or at time of each bronchoscopy (group 2) and assayed for the presence of lymphocyte phenotypes Th1, Th2, Treg, and Th17. After completion of study therapy, patients are followed at 1 month after PDT and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have a diagnosis of non-small cell lung cancer, of any stage, with obstructive or hemorrhagic endobronchial disease receiving PDT treatment.

Exclusion Criteria:

* Patients that have undergone PDT, chemotherapy or radiation therapy within the past 3 months will not be considered for enrollment.
* Patients taking antioxidant therapy will be excluded from enrollment due to potential interaction with the potential oxidative mechanism of action of Photofrin®. These antioxidants would include beta-carotene, lutein, Lycopene, Selenium, Vitamin A, Vitamin C, Vitamin E.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer patients
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Determine the cytokine phenotype found in collected specimens of lung cancer patients treated with photodynamic therapy. | up to one year
  Tumor tissue, broncheoalveolar fluid and blood from enrolled patients will be assayed for the presence of the following defined lymphocyte phenotypes

SECONDARY OUTCOMES:
Correlate the cytokine phenotype of patients undergoing PDT treatment with survival | up to one year
  The immune response that is established will be statistically correlated with the survival rate measured at 6 months and 1 year. This will allow us to discern if a higher survival rate is associated with a specific immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Moffatt-Bruce, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu